CLINICAL TRIAL: NCT00529061
Title: Comprehensive Sickle Cell Centers Collaborative Data Project (C-Data)
Brief Title: Establishing a Database of People With Sickle Cell Disease (Comprehensive Sickle Cell Centers Collaborative Data Project [C-Data])
Acronym: C-Data
Status: Terminated | Type: Observational
Why Stopped: Funds for study ended September 30, 2008.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Susan Lieff, PhD, Rho, Inc. - CSCC Statistics and Data Management Center
Other Study IDs: 1401; U54HL070587-05 (NIH)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-11

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Disease; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause intense pain episodes. The purpose of this study is to gather medical information from children and adults with SCD and establish a database so that researchers can contact people to participate in future SCD research studies.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." The Comprehensive Sickle Cell Centers (CSCC) is a network of 10 centers that conduct research to improve health care and treatment options for people with SCD. This study, the Collaborative Data Project (C-Data), will establish a comprehensive database of children and adults receiving medical care at participating CSCC research centers who are potentially eligible for inclusion in SCD clinical trials. The main purposes of this study are the following: 1) to gather medical information about a large number of people with SCD over a long period of time; 2) to identify potential participants for future SCD clinical trials; 3) to collect information about how SCD affects quality of life; and 4) to evaluate the relationship between SCD patients' characteristics and medical events.

In this study, research staff will review participants' medical records twice a year for at least 5 years. Information will be collected regarding participants' medical history, physical exams, blood tests, and demographics. Once a year, participants will take part in a short interview about their health and lifestyle. Participants will also complete quality-of-life and patient satisfaction questionnaires during the first year of the study and may complete additional questionnaires in the future. During an interview, participants will be asked general questions about their experience with SCD and more specific questions on headaches and any possible relation they may have to SCD pain. Participants may also be asked to provide a blood sample at some point during the study. CSCC researchers will analyze the information in the database and may contact participants in the future to see if they are interested in enrolling in SCD clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD
* Evaluated within the 24 months prior to study entry in the hospital or clinical setting
* Expected to return episodically or regularly for care at one of the CSCCs

Exclusion Criteria:

* Deceased CSCC patient
* Inactive CSCC patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All adult and pediatric patients who have been seen within the last 24 months in the hospital or clinical setting, and are expected to return episodically or regularly for care at one of the CSCCs, are eligible for inclusion in the C-Data project.
Sampling Method: Non-Probability Sample
Enrollment: 3640 (Actual)
Dates: Start 2005-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susi Lieff, PhD, Principal Investigator — Statistics and Data Management Center (SDMC) (RhoFed)
Locations (19):
- United States (19):
  - Children's Hospital of Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Kosair Children's Hospital, Louisville, Kentucky
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital of Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Saint Jude Children's Hospital, Memphis, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - University of Texas Southwestern and Parkland, Dallas, Texas
  - University of Texas at Galveston, Galveston, Texas